CLINICAL TRIAL: NCT00988494
Title: Study of DE-105 Ophthalmic Solution in Patients With Persistent Corneal Epithelial Defect
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01050807
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Persistent Corneal Epithelial Defect

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- High concentration (Experimental): DE-105 high concentration
  Interventions: Drug: DE-105 ophthalmic solution
- Low concentration (Experimental): DE-105 low concentration
  Interventions: Drug: DE-105 ophthalmic solution
- Placebo (Placebo Comparator): DE-105 placebo
  Interventions: Drug: Placebo ophthalmic solution

INTERVENTIONS:
Drug: DE-105 ophthalmic solution — Topical ocular application
  Arms: High concentration
Drug: DE-105 ophthalmic solution — Topical ocular application
  Arms: Low concentration
Drug: Placebo ophthalmic solution — Topical ocular application
  Arms: Placebo

SUMMARY:
Safety and efficacy of DE-105 ophthalmic solution in patients with persistent corneal epithelial defect will be evaluated. Dose-dependent efficacy will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Has corneal epithelial defect and decreased corneal sensitivity.
* Has undergone continuous treatment for corneal epithelial defect for 1 week or longer.

Exclusion Criteria:

* Presence of disease such as active ocular infection, or abnormal lid closure.
* History or presence of chemical burn, Stevens - Johnson Syndrome, etc.
* History of corneal transplantation, LASIK, or hematopoietic stem cell transplantation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-09

PRIMARY OUTCOMES:
Restoration of corneal epithelial defect | Every week

SECONDARY OUTCOMES:
Visual acuity,etc. | Exit visit,etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Japan